CLINICAL TRIAL: NCT05107739
Title: A Phase 1 Safety and Tolerability Study of DeTIL-0255 in Adults With Advanced Malignancies
Brief Title: A Study of DeTIL-0255 in Adults With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Nurix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NX-DeTIL-0255-201
Record Dates: First submitted 2021-10-04; First posted 2021-11-04 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Platinum-resistant Ovarian Cancer; Endometrial Cancer; Cervical Cancer
Keywords: NX-DeTIL-0255; Adoptive Cell Therapy; Tumor Infiltrating Lymphocyte; ACT; TIL; DeTIL
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Run In (Experimental): Patients with gynecological malignancies
  Interventions: Biological: Drug Product De-TIL-0255
- EOC (Experimental): Recurrent or persistent platinum-resistant epithelial ovarian cancer (EOC), including primary peritoneal and fallopian tube carcinoma
  Interventions: Biological: Drug Product De-TIL-0255
- Cervical (Experimental): Recurrent, metastatic, or persistent cervical carcinoma
  Interventions: Biological: Drug Product De-TIL-0255
- Endometrial (Experimental): Advanced or recurrent endometrial cancer
  Interventions: Biological: Drug Product De-TIL-0255

INTERVENTIONS:
Biological: Drug Product De-TIL-0255 — Autologous tumor-infiltrating lymphocytes

SUMMARY:
This is a first-in-human Phase 1 multicenter, open-label oncology study designed to evaluate the safety and efficacy of NX-DeTIL-0255-201 in patients with advanced malignancies.

DETAILED DESCRIPTION:
This study includes a safety run in and a cohort expansion. The safety run in will include patients with any of the indications under study including:

Recurrent or persistent platinum-resistant epithelial ovarian cancer (EOC), including primary peritoneal and fallopian tube carcinoma Recurrent, metastatic, or persistent cervical carcinoma Advanced or recurrent endometrial cancer

Cohort expansion will include patients with advanced malignancies who have received at least two prior systemic therapies in the same indications.

ELIGIBILITY:
Inclusion Criteria:

* One of the following malignancies: Recurrent or persistent platinum-resistant EOC, recurrent, metastatic or persistent carcinoma of the cervix with progression after treatment with taxane-containing regimen, or advance or recurrent endometrial cancer with disease progression after or during second line or greater therapy
* Disease that is metastatic and measurable by RECIST v1.1 criteria
* A resectable lesion for TIL generation
* At least 2 prior lines of therapy
* ≥ 18 years and ≤ 70 years of age
* Life expectancy of at least 4 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ and bone marrow function, in the absence of growth factors
* Patients of child-bearing potential must use adequate contraceptive measures to avoid pregnancy for the duration of the study as defined in the protocol
* A signed consent form indicating that the subjects understands the purpose and procedures required for the study

Exclusion Criteria:

* Known untreated brain metastases
* Uncontrolled intercurrent illness
* History of known seizure disorder
* Unable to comply with study requirements
* Toxicities from previous anticancer therapies that have not resolved to baseline levels or to Grade 1 or less except for alopecia and peripheral neuropathy
* Pregnant, breastfeeding, or planning to become pregnant while enrolled on this study or within 6 months after DeTIL infusion
* Live vaccine within 28 days of first dose of NMA chemotherapy or planned live vaccination within 6 months following DeTIL infusion
* Active known second malignancy with the exception of any of the following: Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or adequately treated follicular or papillary thyroid cancer; or any other cancer from which the patient has been disease-free for ≥ 2 years
* Systemic anti-cancer therapy, including investigational agents, or radiotherapy within 4 weeks of tumor resection
* Major surgery within 4 weeks before tumor resection, or will not have fully recovered from surgery, or has surgery planned within 8 weeks after infusion
* Use of systemic corticosteroids within 15 days (or other immunosuppressive drugs within 30 days) prior to tumor resection
* Use of biotin or other supplements containing higher that the daily adequate intake of biotin
* Clinically significant, uncontrolled cardiac, class III or IV heart failure, thromboembolic events, cardiovascular disease, or history of myocardial infarction within 6 months of planned start of study drug
* History or current evidence of anything that might confound the results of the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 24 Months
  NX-DeTIL-0255-201
Incidence of all deaths | 24 Months
  NX-DeTIL-0255-201
Incidence of dose limiting toxicities | 24 Months
  NX-DeTIL-0255-201
Objective response rate (ORR) per disease-specific response criteria as assessed by the Investigator | 24 Months
  NX-DeTIL-0255-201
Duration of response (DOR) as assessed by the Investigator | 24 Months
  NX-DeTIL-0255-201
Disease control rate (DCR) as assessed by the Investigator | 24 Months
  NX-DeTIL-0255-201
Progression-free survival (PFS) as assessed by the Investigator | 24 Months
  NX-DeTIL-0255-201
Overall survival (OS) as assessed by the Investigator | 24 Months
  NX-DeTIL-0255-201

SECONDARY OUTCOMES:
Changes from baseline in immune cell infiltration in the tumor following DeTIL-0255 infusion | 24 Months
  NX-DeTIL-0255-201

CONTACTS AND LOCATIONS:
Overall Officials: Paula O'Connor, Study Director — Nurix Therapeutics, Inc.
Locations (4):
- United States (4):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No